CLINICAL TRIAL: NCT00226382
Title: Treatment With Peginterferon Alfa-2a (40 KD) (PEGASYS®) of Chronic Hepatitis B Patients, Who Have Failed Anti-viral Treatment. A Pilot Study.
Brief Title: Treatment With Peginterferon Alfa-2a (40 KD) of Chronic Hepatitis B Patients, Who Have Failed Anti-viral Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Professor LY Chan, The Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pegasys Study
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; Pegylated Interferon-alfa-2a; Pegasys
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pegylated Interferon-alfa-2a — Pegasys once weekly

SUMMARY:
This study is to investigate the HBV DNA suppression (and HBeAg seroconversion among HBeAg positive patients) pegylated interferon treatment at 24 weeks after end of treatment among patients who have failed anti-viral treatment in the past.

DETAILED DESCRIPTION:
Chronic hepatitis B is the commonest cause of liver cirrhosis and hepatocellular carcinoma in Hong Kong. Persistent high viraemia and necro-inflammation is associated with higher risk of liver-related complications.

Lamivudine and adefovir dipivoxil are the two anti-viral agents that can suppress the replication of the virus. However, these drugs using either alone or in combination only induce HBeAg seroconversion in less than 20% of patients. Most patients therefore required long-term treatment, which has a risk of development of drug resistance. Premature cessation of these anti-viral agents is usually accompanied by relapse of viraemia and hepatitis.

Pegylated interferon-alfa-2a is modified form of interferon with a 40 kDa polyethylene glycol strand attached to a recombinant interferon. This formulation increases the product's half-life from 7-10 hours to 77 hours. Therefore it can be administered on a more convenient once weekly basis. Pegylated interferon-alfa-2a monotherapy for 24 weeks has been shown to induce sustained HBeAg seroconversion in 35% of patients at the optimal dose of 180 mcg weekly. This drug has been found to be more effective than conventional interferon-alfa in the treatment of chronic hepatitis B as well as chronic hepatitis C.

Data on interferon-based treatment among chronic hepatitis B patients who have failed previous anti-viral treatment is scanty. It is uncertain whether pegylated interferon-alfa-2a treatment will be effective in this group of patients. This is a single-center, pilot study on the virological response of chronic HBV infection to pegylated interferon-alfa-2a among patients who have failed anti-viral treatment in the past. This study will investigate the HBV DNA suppression (and HBeAg seroconversion among HBeAg positive patients) pegylated interferon treatment at 24 weeks after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Positive HBsAg for more than 6 months
* Detectable HBV DNA (patients must have >100,000 copies/ml as measured by PCR)
* HBeAg positive and negative patients are recruited.
* Previous use of nucleoside (nucleotide) analogues for at least 12 months, and the treatment has been stopped for at least 6 months.
* elevated serum ALT > 1.5x upper limited of normal but <= 10X as determined by two abnormal values taken >14 days apart during the six months before the first dose of study drug with at least one of the determinations obtained during the screening period.
* CHB confirmed by liver biopsy in the past or by clinical evaluation.
* Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug. Additionally, all females must be using reliable contraception during the study and for 3 months after treatment completion.

Exclusion Criteria:

* Evidence of decompensated liver disease (Childs B-C), hepato-cellular carcinoma, pre-existing severe depression or other psychiatric disease, significant cardiac disease, significant renal disease, seizure disorders or severe retinopathy.
* Patients who have received antiviral therapy for their chronic hepatitis B or any systemic anti-viral, anti-neoplastic or immuno-modulatory treatment (including supraphysiologic doses of steroids and radiation) within the past 6 months.
* Positive test at screening for anti-HIV, anti-HCV.
* Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation in the study are also excluded. Exception: patients who have had a limited (<=7 days) course of acyclovir for herpetic lesions more than 1 month prior to the first administration of test drug are not excluded.
* Serum total bilirubin > 3X upper limit of normal at screening.
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease.
* History or other evidence of a medical condition associated with chronic liver disease other than HBV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver diseases including Wilson's and alpha1-antitrypsin deficiency, alcoholic liver disease, toxin exposures, thalassemia).
* Women with ongoing pregnancy or who are breast feeding.
* Neutrophil count <1500 cells/mm3 at screening.
* Platelet count <90,000 cells/mm3 at screening.
* Hemoglobin < 11.5 g/dL for females and < 12.5 g/dL for men at screening.
* Serum creatinine level >120 umol/ml for men and >105 umol/ml for women at screening.
* History of severe psychiatric disease, especially depression.
* History of immunologically mediated disease
* History or other evidence of chronic pulmonary disease associated with functional limitation. Severe cardiac disease
* History of a severe seizure disorder or current anticonvulsant use.
* Evidence of an active or suspected cancer or a history of malignancy where the risk of recurrence is > 20% within 2 years. Patients with a lesion suspicious of hepatic malignancy on a screening imaging study will only be eligible if the likelihood of carcinoma is 10% following an appropriate evaluation.
* History of having received any systemic anti-neoplastic (including radiation) or immunomodulatory treatment
* Major organ transplantation.
* Thyroid disease with thyroid function poorly controlled on prescribed medications. Patients with abnormal thyroid stimulating hormone or T4 concentrations, with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease are excluded.
* History or other evidence of severe retinopathy or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
* Patients with a value of alpha-fetoprotein >100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months.
* Evidence of drug and/or alcohol abuse (20g/day for women and 30g/day for men).
* Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening
* Any known history of hypersensitivity to interferon.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
HBeAg positive patients response is defined as HBeAg loss and presence of anti-HBe (HBeAg seroconversion), HBeAg Negative patients response is defined as DNA<20,000 copies/ml and ALT normalization both measured at week 72

SECONDARY OUTCOMES:
Percentage of patients with HBV DNA levels <100,000 copies/ml at week 72, Percentage of patients with HBV DNA levels <10,000 copies/ml at week 72
- Percentage of patients with HBV DNA levels negative by PCR at week 72, ALT normalization at week 72, HBsAg seroconversion at week 72, Safety of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry LY Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Cheng Suen Man Shook Hepatitis Center, Institute of Digestive Disease, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Background] Lai CL, Chien RN, Leung NW, Chang TT, Guan R, Tai DI, Ng KY, Wu PC, Dent JC, Barber J, Stephenson SL, Gray DF. A one-year trial of lamivudine for chronic hepatitis B. Asia Hepatitis Lamivudine Study Group. N Engl J Med. 1998 Jul 9;339(2):61-8. doi: 10.1056/NEJM199807093390201. PMID 9654535
- [Background] Marcellin P, Chang TT, Lim SG, Tong MJ, Sievert W, Shiffman ML, Jeffers L, Goodman Z, Wulfsohn MS, Xiong S, Fry J, Brosgart CL; Adefovir Dipivoxil 437 Study Group. Adefovir dipivoxil for the treatment of hepatitis B e antigen-positive chronic hepatitis B. N Engl J Med. 2003 Feb 27;348(9):808-16. doi: 10.1056/NEJMoa020681. PMID 12606735
- [Background] Leung NW, Lai CL, Chang TT, Guan R, Lee CM, Ng KY, Lim SG, Wu PC, Dent JC, Edmundson S, Condreay LD, Chien RN; Asia Hepatitis Lamivudine Study Group. Extended lamivudine treatment in patients with chronic hepatitis B enhances hepatitis B e antigen seroconversion rates: results after 3 years of therapy. Hepatology. 2001 Jun;33(6):1527-32. doi: 10.1053/jhep.2001.25084. PMID 11391543
- [Background] Cooksley WG, Piratvisuth T, Lee SD, Mahachai V, Chao YC, Tanwandee T, Chutaputti A, Chang WY, Zahm FE, Pluck N. Peginterferon alpha-2a (40 kDa): an advance in the treatment of hepatitis B e antigen-positive chronic hepatitis B. J Viral Hepat. 2003 Jul;10(4):298-305. doi: 10.1046/j.1365-2893.2003.00450.x. PMID 12823597
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Zeuzem S, Feinman SV, Rasenack J, Heathcote EJ, Lai MY, Gane E, O'Grady J, Reichen J, Diago M, Lin A, Hoffman J, Brunda MJ. Peginterferon alfa-2a in patients with chronic hepatitis C. N Engl J Med. 2000 Dec 7;343(23):1666-72. doi: 10.1056/NEJM200012073432301. PMID 11106715
- [Background] Marcellin P, Lau GK, Bonino F, Farci P, Hadziyannis S, Jin R, Lu ZM, Piratvisuth T, Germanidis G, Yurdaydin C, Diago M, Gurel S, Lai MY, Button P, Pluck N; Peginterferon Alfa-2a HBeAg-Negative Chronic Hepatitis B Study Group. Peginterferon alfa-2a alone, lamivudine alone, and the two in combination in patients with HBeAg-negative chronic hepatitis B. N Engl J Med. 2004 Sep 16;351(12):1206-17. doi: 10.1056/NEJMoa040431. PMID 15371578
- [Background] Chan HL, Chui AK, Lau WY, Chan FK, Wong ML, Tse CH, Rao AR, Wong J, Sung JJ. Factors associated with viral breakthrough in lamivudine monoprophylaxis of hepatitis B virus recurrence after liver transplantation. J Med Virol. 2002 Oct;68(2):182-7. doi: 10.1002/jmv.10185. PMID 12210406